CLINICAL TRIAL: NCT01196897
Title: Evaluation of the Next Generation WATCHMAN LAA Closure Technology in Non-Valvular AF Patients
Brief Title: Evaluation of the Next Generation WATCHMAN LAA Closure Technology in Non-Valvular AF Patients (EVOLVE)
Acronym: EVOLVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT1000
Record Dates: First submitted 2010-08-16; First posted 2010-09-09 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2012-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Stroke; Warfarin; Coumadin; TIA; Trans Ischemic Attack
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implantable device (Experimental): WATCHMAN LAA Closure Technology (Gen 4.0)
  Interventions: Device: WATCHMAN LAA Closure Technology (Gen 4.0)

INTERVENTIONS:
Device: WATCHMAN LAA Closure Technology (Gen 4.0) — Implantation of the WATCHMAN device into the left atrial appendage.

SUMMARY:
This study will evaluate the next generation WATCHMAN Left Atrial Appendage (LAA) Closure Device as implanted in patients with non-valvular atrial fibrillation (AF) with a CHADS2 stroke risk stratification score of 1 or greater. This is a prospective, non-randomized study to evaluate the initial use of the next generation WATCHMAN Device.

ELIGIBILITY:
Key Inclusion Criteria:

* Paroxysmal, persistent, or permanent non-valvular atrial fibrillation
* Eligible for long-term Warfarin therapy;
* Eligible to come off Warfarin therapy if the LAA is sealed
* Calculated CHADS2 score of 1 or greater

Key Exclusion Criteria:

* New York Heart Association Class IV Congestive Heart Failure
* Recent MI (within 3 months)
* ASD and/or atrial septal repair or closure device
* Resting heart rate >110 bpm
* Has an implanted mechanical valve prosthesis
* Left atrial appendage is obliterated
* Has undergone heart transplantation
* Has symptomatic carotid disease
* Contraindicated for aspirin
* LVEF < 30%
* Cardiac Tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Successful implantation of the next generation WATCHMAN device without the occurance of life-threatening events caused by the device and/or procedure. | 12-Months
  The implantation of the next generation WATCHMAN device without the occurrence of life-threatening events caused by the device and/or the procedure. These events may include device embolization requiring retrieval, bleeding events such as pericardial effusion requiring drainage, cardiac perforation requiring operation, cranial bleeding events due to any source, and any systemic embolic events related to the device or procedure.
Device Success | Implant through 45-Days
  Device success, defined as successful delivery and release of the WATCHMAN implant into the LAA, including successful re-capture and retrieval if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Na Homolce Hospital
Locations (3):
- NA Homolce Hospital, Prague, Czechia
- Germany (2):
  - Krankenhaus der Barmherzige Bruder, Regensburg, Bavaria
  - Sankt Katharinen Hospital / Cardiovasculares Centrum, Frankfurt